CLINICAL TRIAL: NCT02085148
Title: A Multi-center, Open-label, Non-randomized, Phase I Dose Escalation Study of Regorafenib (BAY 73-4506) in Pediatric Subjects With Solid Malignant Tumors That Are Recurrent or Refractory to Standard Therapy
Brief Title: A Phase I Dose Finding Study in Children With Solid Tumors Recurrent or Refractory to Standard Therapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 15906; 2013-003579-36 (EudraCT Number)
Record Dates: First submitted 2014-03-07; First posted 2014-03-12 (Estimated); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Pediatric Oncology
Keywords: Pediatric cancer; Rhabdomyosarcoma,; Ewing sarcoma; Hepatoblastoma; Neuroblastoma; Wilm's tumor
MeSH Terms: conditions — Neoplasms; Rhabdomyosarcoma; Sarcoma, Ewing; Hepatoblastoma; Neuroblastoma; Wilms Tumor | interventions — regorafenib; Vincristine; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sequential dosing schedule (Experimental): Expansion phase: Schedule B - Sequential dosing schedule: Of a 21-day cycle, regorafenib will be dosed sequentially, following administration of VI: Vincristine：intravenous bolus, 1.5 mg/m2 (0.05 mg/kg for subjects ≤ 10 kg), Day 1 and Day 8. Irinotecan: intravenously over 1 hour, 50mg/m2/day, Day 1 to Day 5. Regorafenib: orally, at a starting dose level of 72 mg/m2 (subjects 2 to less than 18 years old) or 60 mg/m2 (subjects 6 to less than 24 months old) once daily, Day 8 to Day 21.
  Interventions: Drug: Regorafenib (BAY73-4506); Drug: Vincristine (Cellcristin®); Drug: Irinotecan (Irinotecan Cell pharm®)
- Concomitant dosing schedule (Experimental): Expansion phase: Schedule A - Concomitant dosing schedule: Of a 21-day cycle, regorafenib will be concomitantly administered with vincristine and irinotecan (VI): Vincristine: intravenous bolus, 1.5 mg/m2 (0.05 mg/kg for subjects ≤ 10 kg), Day 1 and Day 8. Irinotecan: intravenously over 1 hour, 50 mg/m2/day, Day 1 to Day 5. Regorafenib: orally, at a starting dose level of 72 mg/m2 (subjects 2 to less than 18 years old) or 60 mg/m2 (subjects 6 to less than 24 months old) once daily, Day 1 to Day 14.
  Interventions: Drug: Regorafenib (BAY73-4506); Drug: Vincristine (Cellcristin®); Drug: Irinotecan (Irinotecan Cell pharm®)
- Dose escalation (Experimental): Dose escalation phase: This phase of the study has been completed
  Interventions: Drug: Regorafenib (BAY73-4506)

INTERVENTIONS:
Drug: Regorafenib (BAY73-4506) — Regorafenib will be given orally once a day, across cycles of 21 days each. During each cycle regorafenib is taken for 2 weeks followed by one week off the drug. Doses of the study drug used in this study are age-dependent and the children's dose will been adjusted based on the age and the body surface area and given either as tablets or granulate.
Drug: Vincristine (Cellcristin®) — Vincristine will be given at a dose of 1.5 mg/m2 (0.05 mg/kg for subjects ≤ 10 kg, maximum 2.0 mg) on Day 1 and Day 8 in 21-day cycles.
  Arms: Concomitant dosing schedule; Sequential dosing schedule
Drug: Irinotecan (Irinotecan Cell pharm®) — Irinotecan will be administered at a starting dose of 50 mg/m2/day from Day 1 to Day 5, in 21 day cycles.
  Arms: Concomitant dosing schedule; Sequential dosing schedule

SUMMARY:
Dose escalation phase of the study :

To define the safety profile, maximum tolerated dose (MTD) and recommended phase II dose (RP2D) of regorafenib administered orally as a single agent in a 3-weeks-on/1- week-off schedule in repeating cycles of 28 days in pediatric subjects with solid malignant tumors recurrent or refractory to standard therapy. To characterize the pharmacokinetics (PK) of regorafenib The dose escalation phase of the study has been completed.

Expansion phase:

To define the safety profile, MTD and the RP2D of regorafenib administered orally in combination with backbone chemotherapy (vincristine and irinotecan) at relapse in pediatric subjects with rhabdomyosarcoma (RMS) and other solid malignant tumors recurrent or refractory to standard therapy.

DETAILED DESCRIPTION:
Expansion Phase of the study:

Subjects must have relapsed/refractory RMS or a solid malignant tumor (Ewing sarcoma, hepatoblastoma, neuroblastoma and Wilms tumor).

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form by subjects and/or subjects' parents/legal guardians and age appropriate Assent Form by the subjects obtained before any study specific procedure
* Age: from 6 months to less than 18 years old
* Diagnosis, Dose escalation phase of the study: subjects must have had histologic verification of solid malignancy at original diagnosis. Subjects with recurrent or refractory solid tumors are eligible, including primary central nervous system (CNS) tumors or subjects with known CNS metastases. Subject's current disease state must be one for which there is no known effective therapy or therapy proven to prolong survival with an acceptable quality of life. Effective therapy may include surgery, radiation therapy, chemotherapy or any combination of these modalities.

Dose expansion phase of the study: subjects must have relapsed/refractory RMS or a solid malignant tumor (Ewing sarcoma, hepatoblastoma, neuroblastoma and Wilms tumor) in which treatment with vincristine/irinotecan is considered backbone chemotherapy at relapse and a scientific rationale to combine vincristine/irinotecan with regorafenib exists.

* Subjects must have at least one measurable or evaluable lesion according to Response Evaluation Criteria in Solid Tumors (RECIST), version 1.1. For the neuroblastoma subjects with osteomedullary disease, the SIOPEN (International Society of Pediatric Oncology Europe Neuroblastoma Group) score will be used. Bone scans (if clinically indicated) should be obtained ≤12 weeks prior to the start of treatment.
* Life expectancy of at least 12 weeks from the time of signing informed consent/assent.
* Performance level: Karnofsky ≥ 70% for subjects > 12 years of age or Lansky ≥ 70% for subjects ≤ 12 years of age
* Adequate hematological function assessed by the following laboratory requirements conducted within 7 days before starting study treatment:

Peripheral absolute neutrophil count (ANC): ≥ 1.0 x 10*9/L Platelet count : ≥ 100 x 10*9/L (transfusion independent) Hemoglobin: ≥ 8.0 g/dL

-Adequate hepatic function defined as:

* Aspartate aminotransferase/alanine aminotransferase (AST/ALT) ≤ 3.0* ULN
* Bilirubin (sum of conjugated and unconjugated) ≤ 1.5 * ULN

Exclusion Criteria:

* Prior treatment with regorafenib. Subjects permanently withdrawn from study participation will not be allowed to re-enter the study.
* Dose expansion phase of the study only: Subjects with brain tumors or subjects with known CNS metastases are excluded.
* Subjects with uncontrolled baseline hypertension higher than Grade 1 NCICTCAE v. 4.0
* Subjects with evidence or history of disorders of coagulation or thrombosis
* Cardiac abnormalities and cardiac arrhythmias requiring anti-arrhythmic therapy (beta blockers or digoxin are permitted)
* History of organ allograft (including allogeneic bone marrow transplant)
* Any other malignant disease treated prior to study entry
* Pregnancy or breast feeding
* Significant gastrointestinal disorders with diarrhea as a major symptom e.g., Crohn's disease or any malabsorption condition
* Close affiliation with the investigational site, e.g. a close relative of the investigator or a dependent person (e.g. employee or student of the investigational site)
* Unresolved toxicity higher than NCI-CTCAE v. 4.0 Grade 1 attributed to any prior therapy/procedure (excluding alopecia, chemotherapy-induced ototoxicity, Grade 2 chemotherapy-induced neuropathy and, as per above eligibility criteria, anemia with hemoglobin ≥ 8 mg/dL and ANC ≥ 1.0 x 10 9/L ).
* Any other malignant disease treated prior to the study

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 62 (Actual)
Dates: Start 2014-04-11 (Actual); Primary Completion 2019-05-05 (Actual); Study Completion 2024-03-13 (Actual)

PRIMARY OUTCOMES:
Safety: Maximum Tolerated Dose | approximately after 21 months
  MTD is defined as the dose level at which none or 1 of 6 participants experiences dose-limiting toxicity (DLT), when at least 2 of 3-6 participants experience a DLT at the next highest dose
Safety: Recommended Phase II Dose | approximately after 21 months
  In order to establish a RP2D, the MTD cohort will be expanded to have at least 12 evaluable subjects to confirm the RP2D. It is expected that at least 15 subjects evaluable for DLTs will be necessary to establish the RP2D of the combination"
Number of participants with Adverse Events | Dose escalation phase:approximately after 21 months; Expansion Phase: approximately after 21 months
  Individual listings of adverse events will be provided. The incidence of treatment-emergent adverse events and drug-related adverse events, respectively, will be summarized by worst NCI-CTCAE v 4.0 grade and by dose level
AUC(0-24)md based on nominal dosing | Dose escalation phase:Cycle 1 Day 1, Day 15 and Day 21
  Dose escalation phase has been completed

SECONDARY OUTCOMES:
Overall survival | Dose escalation phase: approximately 21 months; Expansion phase: approximately 21 months
Time to progression | Dose escalation phase: approximately 21 months; Expansion phase: approximately 21 months
Tumor response: tumor assessment by RECIST v. 1.1 | Dose escalation phase: approximately 21 months; Expansion phase: approximately 21 months
Taste and texture questionnaire of the regorafenib formulations | Dose escalation phase: Cycle 1; Expansion phase:Concomitant: Cycle 1 Day 1;Sequential: Cycle 1 Day 8
  Expansion phase Dose escalation phase
AUC(0-24)md based on nominal dosing | Expansion Phase:Cycle 1 Day1, Day 15 and Day 21
  Expansion phase
Cmax(0-24)md based on individual dosing | Expansion Phase:Cycle 1 Day1, Day 15 and Day 21
  Expansion phase
Cav(0-24)md based on individual dosing | Expansion phase:Cycle 1 Day1, Day 15 and Day 21; Dose escalation phase:Cycle 1 Day1, Day 15 and Day 21
  Expansion phase Dose escalation phase
t1/2eff,md based on individual dosing | Expansion phase:Cycle 1 Day1, Day 15 and Day 21; Dose escalation phase:Cycle 1 Day1, Day 15 and Day 21
  Expansion phase Dose escalation phase
AUC(0-24)md based on individual dosing | Expansion Phase:Cycle 1 Day1, Day 15 and Day 21
  Expansion phase
Clearance of irinotecan and SN-38 | Expansion Phase:Cycle 1 Day1, Day 15 and Day 21
  Expansion phase

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (12):
- France (4):
  - Lyon
  - Marseille
  - Paris
  - Villejuif
- Italy (2):
  - Genoa, Liguria
  - Milan, Lombardy
- Spain (2):
  - Madrid
  - Valencia
- United Kingdom (4):
  - Sutton, Surrey
  - Newcastle upon Tyne, Tyne and Wear
  - Birmingham, West Midlands
  - Manchester

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

REFERENCES:
- [Derived] Casanova M, Bautista F, Campbell-Hewson Q, Makin G, Marshall LV, Verschuur AC, Canete Nieto A, Corradini N, Ploeger BA, Brennan BJ, Mueller U, Zebger-Gong H, Chung JW, Geoerger B. Regorafenib plus Vincristine and Irinotecan in Pediatric Patients with Recurrent/Refractory Solid Tumors: An Innovative Therapy for Children with Cancer Study. Clin Cancer Res. 2023 Nov 1;29(21):4341-4351. doi: 10.1158/1078-0432.CCR-23-0257. PMID 37606641
- [Derived] Geoerger B, Morland B, Jimenez I, Frappaz D, Pearson ADJ, Vassal G, Maeda P, Kincaide J, Mueller U, Schlief S, Teufel M, Ploeger BA, Cleton A, Agostinho AC, Marshall LV. Phase 1 dose-escalation and pharmacokinetic study of regorafenib in paediatric patients with recurrent or refractory solid malignancies. Eur J Cancer. 2021 Aug;153:142-152. doi: 10.1016/j.ejca.2021.05.023. Epub 2021 Jun 20. PMID 34157616